CLINICAL TRIAL: NCT02455193
Title: Neuronal Effects of Exercise in Schizophrenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14-1282; UL1TR001082 (NIH); R01MH102224 (NIH)
Record Dates: First submitted 2015-05-21; First posted 2015-05-27 (Estimated); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Exercise; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise intervention (Experimental): 10 weeks of a moderate exercise intervention
  Interventions: Behavioral: Exercise
- Diet intervention (Active Comparator): 10 weeks of a diet intervention
  Interventions: Behavioral: Diet

INTERVENTIONS:
Behavioral: Exercise
  Arms: Exercise intervention
Behavioral: Diet
  Arms: Diet intervention

SUMMARY:
This study plans to learn more about how common drugs prescribed to individuals with schizophrenia contribute to weight gain, as well as how exercise and diet impact appetite and the brain's response to food. In this study, the investigators will be evaluating how participants' brains respond to food images as well as asking questions about their food preferences and intake and clinical symptoms. The investigators may also ask participants to complete an exercise or diet intervention to see how this changes brain responses or food preferences.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder
* Between 21 and 70 years of age
* Currently prescribed either olanzapine, risperidone, clozapine, or haloperidol, OR not currently being treated with any neuroleptic medications
* Weight stable within 5 percent for the last 6 months

Exclusion Criteria:

* Pregnancy
* Substance abuse
* Significant endocrine/metabolic disease (e.g., uncontrolled hypertension, severe hypertriglyceridemia)
* MRI-specific exclusion criteria (e.g., claustrophobia, metal in the body)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-08; Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Neuronal response to visual food cues | 14 weeks
  Neuronal response (insula) while viewing visual food cues
Resting-state neuronal response | 14 weeks
  Neuronal response (default mode network) during rest

SECONDARY OUTCOMES:
Appetite Rating on a visual analogue scale (VAS) | 14 weeks
  Participants will be asked to rate their hunger via Hunger ratings on a VAS
Fasting leptin | 14 weeks
  Fasting blood levels of leptin
Fasting ghrelin | 14 weeks
  Fasting blood levels of ghrelin

CONTACTS AND LOCATIONS:
Overall Officials: Jason Tregellas, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No